CLINICAL TRIAL: NCT01779635
Title: Continuous Renal Replacement Therapy With Anticoagulation-free Regimen in Bleeding-risk Patients Using oXiris Membrane - CARROM Study
Brief Title: Efficacy and Safety of Heparin-grafted Membrane for CRRT
Acronym: CARROM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: DSRB 2012/02222; NKFRC/2012/01/11 (Other Grant/Funding Number: National Kidney Foundation Singapore)
Record Dates: First submitted 2013-01-27; First posted 2013-01-30 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Acute Kidney Injury; Hemorrhage; Coagulopathy
Keywords: Heparin-grafted membrane; Circuit lifespan; Continuous renal replacement therapy; Anticoagulation free; Bleeding risk; Acute kidney injury; Critical illness
MeSH Terms: conditions — Acute Kidney Injury; Hemorrhage; Hemostatic Disorders; Critical Illness

STUDY DESIGN:
Intervention Model Description: Randomized initiation with oXiris versus M150 (conventional filter), with cross-over for subsequent circuits.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oXiris as first filter (Active Comparator): Start off the first CRRT circuit with oXiris, then cross-over to M150, then oXiris, then back to M150
  Interventions: Device: oXiris as first filter
- M150 as first filter (Other): Patients in M150 arm will start off with M150 as first filter for CRRT, then cross-over to oXiris after the former clots, then back to M150, then to oXiris.
  Interventions: Device: M150 as first filter

INTERVENTIONS:
Device: oXiris as first filter — 2 arms - each start off CRRT with either oXiris or M150 as first hemofilter, and then do cross-over to either hemofilters in a sequential manner when the former clots
  Arms: oXiris as first filter
Device: M150 as first filter — start off with M150 as first hemofilter, then cross-over to oXiris when former clots, and then to M150, and then lastly to oXiris
  Arms: M150 as first filter

SUMMARY:
The investigators hypothesize that the use of heparin-grafted membrane versus conventional membrane in critically-ill patients with bleeding-risk undergoing continuous renal replacement therapy, will effectively prolong the circuit lifespan, without worsening of the systemic APTT or underlying bleeding risk.

DETAILED DESCRIPTION:
Aims and objectives:

We aim to compare the performance and safety of heparin-grafted AN69 membrane (oXiris, Gambro) with the conventional AN69 membrane (M150, Gambro) without systemic anticoagulation during continuous renal replacement therapy (CRRT), in critically ill patients with acute kidney injury (AKI) admitted to the intensive care unit (ICU), who has moderate bleeding risk and in whom systemic anticoagulation is contraindicated.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (age 21 and above) who are admitted to ICUs or CCU and requiring CRRT for acute kidney injury or ESRD Patients who has moderate bleeding risk (see below definitions) Patients with NO systemic or regional circuit anticoagulation Informed consent taken from the patient, or proxy if the former is unable to sign due to medical reasons Anticipated need for prolonged CRRT > 3 days

(Moderate bleeding risk criteria:)

Moderate bleeding risk is defined by any of the following:

1. Platelet count < 100 x 109 mm3 (but > 50)
2. INR > 1.5 (but < 2.5)
3. APTT > 50 seconds (but < 75)
4. Post-surgery for < 48 hours
5. Post-invasive procedures (eg. Pericardiocentasis) < 24 hrs
6. Post major artery puncture or catheter removal from major arteries (carotids, subclavian, or femoral) < 24 hours
7. Recent internal or gastrointestinal bleeding within 48 hours (should be secured bleeding with no relapse noted)

Exclusion Criteria:

Patients with very high bleeding risk (for which they should also fall outside of the below inclusion criteria - see below) Patients who are known to have heparin-induced thrombocytopenia or allergic to heparin Patients with other medical conditions for which heparin is contraindicated. Patients who require systemic anticoagulation for medical indications (We will accept patients who are on prophylactic doses of anticoagulation for DVT prophylaxis) Patients who are pregnant Patients/legally accepted surrogate who decline to consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Circuit lifespan during continuous renal replacement therapy (up till termination as defined above) with each dialyzer (oXiris or M150) | usually 10 - 30 hours from commencement of circuit
  Circuit lifespan

SECONDARY OUTCOMES:
Pre-circuit INR/APTT, and post-circuit INR/APTT 2 hours after termination. (We will be using the 2 hour post-circuit APTT result of the preceding dialyzer, as the pre-circuit APTT for the subsequent dialyzer. | Usually after 10-30 hours when dialyzer clots
  effect on coagulation status
Serum urea/creatinine, and effluent urea/creatinine (paired samples) at 4 hrs from each circuit commencement, to examine "protein layering" and solute clearance. | Usually 4 hours into circuit commencement
  effect on clearance
Transmembrane pressure (TMP), pressure drop across hemodiafilter (PDF), pressure in (PI), will be recorded on hourly basis throughout treatment, as per usual nursing protocol. | over 10-30 hours of circuit running
  effect on circuit pressures

OTHER OUTCOMES:
Total inotropic score, which is defined as total quantities of Dopamine + Dobutamine + 100 (Noradrenaline) + 100 (Adrenaline) in mcg/kg/min; pre- and post- use of the circuit. | usually after 10-30 hours of circuit lifespan
  effect on hemodynamics
Urine output over the 6 hours preceding the commencement of first circuit, and 6 hours after termination of the first circuit. | Usually after 10-30 hours of circuit lifespan
  effect on oliguria

CONTACTS AND LOCATIONS:
Overall Officials: Horng-Ruey Chua, MBBS, Principal Investigator — National University Health System
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schetz M, Van Cromphaut S, Dubois J, Van den Berghe G. Does the surface-treated AN69 membrane prolong filter survival in CRRT without anticoagulation? Intensive Care Med. 2012 Nov;38(11):1818-25. doi: 10.1007/s00134-012-2633-x. Epub 2012 Jul 7. PMID 22773036
- [Background] Uchino S, Fealy N, Baldwin I, Morimatsu H, Bellomo R. Continuous is not continuous: the incidence and impact of circuit "down-time" on uraemic control during continuous veno-venous haemofiltration. Intensive Care Med. 2003 Apr;29(4):575-8. doi: 10.1007/s00134-003-1672-8. Epub 2003 Feb 8. PMID 12577144
- [Background] Evenepoel P, Dejagere T, Verhamme P, Claes K, Kuypers D, Bammens B, Vanrenterghem Y. Heparin-coated polyacrylonitrile membrane versus regional citrate anticoagulation: a prospective randomized study of 2 anticoagulation strategies in patients at risk of bleeding. Am J Kidney Dis. 2007 May;49(5):642-9. doi: 10.1053/j.ajkd.2007.02.001. PMID 17472846
- [Background] Tan HK, Baldwin I, Bellomo R. Continuous veno-venous hemofiltration without anticoagulation in high-risk patients. Intensive Care Med. 2000 Nov;26(11):1652-7. doi: 10.1007/s001340000691. PMID 11193272
- [Background] Chua HR, Baldwin I, Bailey M, Subramaniam A, Bellomo R. Circuit lifespan during continuous renal replacement therapy for combined liver and kidney failure. J Crit Care. 2012 Dec;27(6):744.e7-15. doi: 10.1016/j.jcrc.2012.08.016. Epub 2012 Oct 24. PMID 23102533
- [Derived] Tsujimoto Y, Miki S, Shimada H, Tsujimoto H, Yasuda H, Kataoka Y, Fujii T. Non-pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2021 Sep 14;9(9):CD013330. doi: 10.1002/14651858.CD013330.pub2. PMID 34519356